CLINICAL TRIAL: NCT06434818
Title: Development and Evaluation of Enhanced Digital-Chemosensory-Based Olfactory Training for Remote Management of Substance Use Disorders (EDITOR)
Brief Title: Enhanced Digital-Chemosensory-Based Olfactory Training for Remote Management of Substance Use Disorders
Acronym: EDITOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Evon Medics LLC (Industry)
Collaborators: Howard University (Other); Maryland Treatment Center (Unknown); Clinics of Dr. Edwin Chapman, MD, PC @ MHDG (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDITDA056156; 4R44DA056156-02 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Substance Use Disorders; Opioid Use Disorder; Alcohol Use Disorder; Cocaine Use Disorder; Methamphetamine-dependence
Keywords: Substance Abuse; Substance Use Disorder; Retention; Relapse; Chemosensory-Based Olfactory Networks Training; Remote Management
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Alcoholism; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Enhanced Digital-Chemosensory-Based Olfactory Training (EDITOR) (Experimental): The EDITOR device is designed to stimulate intensive neural activity in OFC over long periods of time. It consists of 40 daily cycles of intervention with a combination of olfactory stimulation and training tasks, lasting ~45 minutes, delivered once daily over three months. The device also includes 60% beta-caryophyllene chemosensory stimulation to target AUD and stimulant use disorder and 10 digital enhancements for the purpose of remote treatment, remote acquisition of behavioral and physiological data, and seamless data transmission to providers, through a HIPAA-compliant clinic end portal.
  Participants assigned to this arm will receive their treatment-as-usual (TAU) alongside daily EDITOR therapy for three months. TAU will depend on the drug abused [Buprenorphine with a median dose of 24 mg (range 16 - 32 mg) for Opioid use disorder and naltrexone (50-100 mg daily for Alcohol use disorder (AUD).
  Interventions: Combination Product: EDITOR (CBOT with olfactory stimulants, OFC tasks & remote monitoring of treatment compliance)
- Chemosensory-Based Olfactory Training (CBOT) (Active Comparator): CBOT with olfactory stimulants & orbitofrontal (OFC) tasks
  TAU same as above + CBOT (Chemosensory-Based Olfactory Training) therapy (40 cycles of olfactory stimulation and OFC training tasks, lasting ~45 minutes, once daily over three months) + use of their smartphone to communicate with their clinic provider/staff
  Interventions: Combination Product: CBOT with olfactory stimulants & OFC tasks
- Chemosensory-Based Olfactory Training (CBOT) Sham (Sham Comparator): Control Device (Sham) is CBOT device without olfactory stimulants and orbitofrontal tasks.
  TAU same as above + CBOT sham + use of their smartphone to communicate with their clinic provider/staff. This CBOT device uses compressed room air scented with phenylethylamine (rose scent) instead of olfactory stimulants and has shape pattern matching tasks instead of cognitive tasks in order to blind users to their treatment assignment. Similar to the active arm, sham COT will be used daily for 45 minutes.
  Interventions: Combination Product: CBOT Sham

INTERVENTIONS:
Combination Product: EDITOR (CBOT with olfactory stimulants, OFC tasks & remote monitoring of treatment compliance) — EDITOR includes a user-friendly cloud portal synced with the main device, providing a comprehensive training program for the orbitofrontal cortex (OFC). The main device stimulates the orbitofrontal cortex intensely, preventing habituation to smells and improving adaptability. This enhances neurobehavioral plasticity, benefiting Substance Use Disorder (SUD) outcomes. The device also features a 60% beta-caryophyllene scent for addressing issues like Alcohol Use Disorder and stimulant use disorders. With ten digital enhancements, it enables remote treatment and data collection, seamlessly transmitting information to healthcare providers through a secure, HIPAA-compliant portal.
  Other Names: EDITOR plus Treatment-As-Usual (TAU)
  Arms: Enhanced Digital-Chemosensory-Based Olfactory Training (EDITOR)
Combination Product: CBOT with olfactory stimulants & OFC tasks — The CBOT with proprietary odorant molecules is designed to stimulate olfactory neural activity over long periods of time combined with orbitofrontal cortex (OFC) dependent olfactory tasks.
  Other Names: CBOT active plus TAU
  Arms: Chemosensory-Based Olfactory Training (CBOT)
Combination Product: CBOT Sham — CBOT Sham uses artificially scented compressed room air instead of olfactory stimulants and has control cognitive olfactory tasks
  Other Names: CBOT passive plus TAU
  Arms: Chemosensory-Based Olfactory Training (CBOT) Sham

SUMMARY:
The overarching goal of this study phase, Phase II component is to implement Enhanced Digital-Chemosensory-Based Olfactory Training for Remote Management of Substance Use Disorders (EDITOR) device in substance use disorder (SUD) clinics to demonstrate pilot effectiveness for SUD outcomes compared to treatment as usual (TAU) and Computerized Chemosensory-Based Orbitofrontal Networks Training (CBOT) device as active control. The investigators will conduct a multi-site study of 300 adult patients with opiate use disorder (OUD), stimulant (i.e., cocaine, methamphetamine) and/or alcohol use disorder (AUD) from community and clinics to evaluate whether EDITOR is associated with better patient treatment outcomes (e.g., retention in treatment and abstinence). The pilot study will provide preliminary data needed for design of a Phase III trial, including estimates of effect size. The investigators will also explore development of machine learning/AI algorithms integrating clinical and physiological data into treatment decision guides for providers.

DETAILED DESCRIPTION:
The Development and Evaluation of Enhanced Digital-Chemosensory-Based Olfactory Training for Remote Management of Substance Use Disorders (EDITOR) is a project to develop a sustainable, scalable, and patient-centered mobile health platform, comprised of (1) a patient-facing culturally-adapted digital chemosensory therapeutic for stimulant, alcohol and opioid use disorders, sensors for acquisition of objective physiological measures of substance intoxication and withdrawal, and an application for running and interpreting the interventions and sensory acquisition programs; and (2) a provider-facing web portal, for substance use disorder treatment in socially disadvantaged and sexual minority populations.

The small business, Evon Medics implemented the use of the EDITOR device as a novel approach for remote management of substance use disorders (SUDs) amid the challenges of the COVID-19 pandemic. Management of SUD mostly involve direct contact between patients and providers, but the precedence of COVID-19 pandemic has elevated the need for patient-centered remote management of SUD. While digital therapeutics and mobile health platforms provide avenues for remote management, communities of African Americans (AA), Hispanic Americans (HA) and other socially disadvantaged populations lag in adoption of these mobile platforms, due to inability to read, digital illiteracy, lack of access to smartphones, absence of reliable Wi-Fi or internet, and financial constraints. Moreover, while interventions exist for OUD, there are no drugs for cocaine or stimulant use disorders. Underserved AA and HA communities with OUD, particularly marginalized men who have sex with men (MSM), have more severe co-existing cocaine, methamphetamine, and alcohol use disorders; and digital solutions for these populations are lacking. Providers on the other hand, lack well-adapted, intelligent-based physiological and psychophysical acquisition platforms to guide remote agonist management of opioid and alcohol withdrawal.

EVON Medics developed a combinatorial digital chemosensory-based orbitofrontal cortex training for Opioid Use Disorder (CBOT). Based on the limitations of CBOT for the socially disadvantaged AA, HA and MSM population, the investigators recently revised the platform for treatment of stimulant and alcohol use disorder, by including beta-caryophyllene chemosensory stimulation. Further product development, with innovative changes to the patient-facing platform and a new provider-facing platform to guide remote management of OUD, stimulant (cocaine and methamphetamine) use and alcohol use disorders were preliminary tested (Phase I) in affiliated substance use community programs and community populations in the under-served communities in Washington, DC and Maryland.

In this study phase, Phase II of this Fast-Track SBIR application, the investigators will conduct a pilot randomized trial of EDITOR compared to treatment as usual and CBOT for office-based treatment of SUDs in several federal funded programs associated with Evon Medics and Howard University, to assess EDITOR's effectiveness in improving treatment retention, reducing relapses, and mitigating SUD severity, and offering a promising solution for home-based SUD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 years, inclusive at enrollment.
2. Diagnosis of current moderate or severe substance use disorders, opioid use disorders, stimulant (cocaine and methamphetamine) use, and alcohol use disorders in the past three months, including the past month.
3. Does not meet criteria for other current SUDs outside of the 3 above, except for mild or moderate use of cannabis
4. Willing to receive study interventions and buprenorphine (for OUD group) and naltrexone (for AUD group) during the study
5. Females must not be pregnant at enrollment and agree not to become pregnant during the trial, through scientifically valid ways of contraception
6. Willing to sign the informed consent form.
7. Have a stable place to stay and retain the EDITOR devices in a secure condition when receiving the intervention and during the entire duration of the study participation.

Exclusion Criteria:

1. Any significant neurological disease such as stroke, dementia, meningitis, neurosyphilis, cerebral palsy, encephalitis, epilepsy, or seizures.
2. Mental retardation.
3. Presence of serious mental illness, such as schizophrenia, bipolar disorders, and suicidal risk. Diagnosis of major depressive disorders, anxiety disorders, and post-traumatic stress disorders (PTSD), will be included if symptoms are stable, with no suicidal ideas or plans, and there are no recent changes in treatment of these conditions in the 6 weeks prior to enrollment.
4. Experiencing current suicide ideas or plans.
5. Any unstable medical condition such as uncontrolled hypertension, uncontrolled diabetes, or liver cirrhosis as determined by the site PI.
6. History of severe traumatic nose injury that affects the ability to smell or significant intranasal disease, as determined by the site PI.
7. Known allergies or intolerance to aromas from plant essential oils. E.g., orange and lemon.
8. Breastfeeding or pregnancy test positive or plans to get pregnant in the 6 months following enrollment.
9. Individuals who are on parole or probation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Retention in SUD treatment | Baseline to day 14
  3-month retention in SUD treatment, is defined as missing two consecutive clinic visits after completing the first two weeks of SUD treatment; the rationale is to allow for buprenorphine (BUP) dose stabilization in those with opiate use disorder (OUD). Investigators found that missing two visits strongly correlated with self-reported relapse, positive drug urine screen, and non-adherence to the buprenorphine.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
Retention in SUD treatment | Baseline to day 28
  3-month retention in SUD treatment, is defined as missing two consecutive clinic visits after completing the first two weeks of SUD treatment; the rationale is to allow for buprenorphine (BUP) dose stabilization in those with opiate use disorder (OUD). Investigators found that missing two visits strongly correlated with self-reported relapse, positive drug urine screen, and non-adherence to the buprenorphine.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
Retention in SUD treatment | Baseline to 8 weeks
  3-month retention in SUD treatment, is defined as missing two consecutive clinic visits after completing the first two weeks of SUD treatment; the rationale is to allow for buprenorphine (BUP) dose stabilization in those with opiate use disorder (OUD). Investigators found that missing two visits strongly correlated with self-reported relapse, positive drug urine screen, and non-adherence to the buprenorphine.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
Retention in SUD treatment | Baseline to three months
  3-month retention in SUD treatment, is defined as missing two consecutive clinic visits after completing the first two weeks of SUD treatment; the rationale is to allow for buprenorphine (BUP) dose stabilization in those with opiate use disorder (OUD). Investigators found that missing two visits strongly correlated with self-reported relapse, positive drug urine screen, and non-adherence to the buprenorphine.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
SUD Relapse Rate | Baseline to day 7
  Relapse is defined as presence of self-reported repeat (i.e., 2 or more) specific substance use after the first week, and/or presence of positive urine drug test for opiates.
  Ascertainment of relapse is through:
  1. survey question administered weekly, inquiring how many days in the past 1 week did the subject use drugs or alcohol; the dates of substance use; and the quantity (or dose) of drugs used; and
  2. biochemical verification of drug use from urine samples collected and tested every two weeks.
SUD Relapse Rate | Baseline to day 14
  Relapse is defined as presence of self-reported repeat (i.e., 2 or more) specific substance use after the first week, and/or presence of positive urine drug test for opiates.
  Ascertainment of relapse is through:
  1. survey question administered weekly, inquiring how many days in the past 1 week did the subject use drugs or alcohol; the dates of substance use; and the quantity (or dose) of drugs used; and
  2. biochemical verification of drug use from urine samples collected and tested every two weeks.
SUD Relapse Rate | Baseline to day 28
  Relapse is defined as presence of self-reported repeat (i.e., 2 or more) specific substance use after the first week, and/or presence of positive urine drug test for opiates.
  Ascertainment of relapse is through:
  1. survey question administered weekly, inquiring how many days in the past 1 week did the subject use drugs or alcohol; the dates of substance use; and the quantity (or dose) of drugs used; and
  2. biochemical verification of drug use from urine samples collected and tested every two weeks.
SUD Relapse Rate | Baseline to 8 weeks
  Relapse is defined as presence of self-reported repeat (i.e., 2 or more) specific substance use after the first week, and/or presence of positive urine drug test for opiates.
  Ascertainment of relapse is through:
  1. survey question administered weekly, inquiring how many days in the past 1 week did the subject use drugs or alcohol; the dates of substance use; and the quantity (or dose) of drugs used; and
  2. biochemical verification of drug use from urine samples collected and tested every two weeks.
SUD Relapse Rate | Baseline to three months
  Relapse is defined as presence of self-reported repeat (i.e., 2 or more) specific substance use after the first week, and/or presence of positive urine drug test for opiates.
  Ascertainment of relapse is through:
  1. survey question administered weekly, inquiring how many days in the past 1 week did the subject use drugs or alcohol; the dates of substance use; and the quantity (or dose) of drugs used; and
  2. biochemical verification of drug use from urine samples collected and tested every two weeks.
SUD engagement | Baseline to day 14
  SUD engagement is the proportion of people treated at baseline who complete the first two weeks of treatment.

SECONDARY OUTCOMES:
Opioid Craving Scale (OCS) | Baseline to Day 7
  Change in pre- and post- intervention changes using OCS
  The Opioid Craving Scale is used to measure opioid craving. The scale consists of three items rated on a visual analogue scale from 0-10: (1) How much do you currently crave opiates? (rated from not at all to extremely), (2) In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates (rated from no desire to extremely strong), and (3) Please imagine yourself in the environment in which you previously used opiates. If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today? (rated from not at all to I'm sure I would use opiates).
Cocaine Craving Questionnaire-Brief (CCQ-Brief) | Baseline to day 7
  Change in pre- and post- intervention changes using CCQ-Brief
  The Cocaine Craving Questionnaire-Brief (CCQ-Brief) consists of 10 statements about the respondent's feelings and thoughts about using cocaine as her or she is completing the questionnaire (i.e., right now). This instrument allows investigators to obtain a reflection of the respondent's general cocaine craving.
Self-report instruments for Alcohol Craving | Baseline to day 7
  Change in pre- and post- intervention changes using self-report instruments for alcohol craving
  Administration of a single-item instrument on which the participant reports his or her level of subjective craving. These instruments include questions such as "How strong is your craving for alcohol?" or "How strong is your urge to drink?"
Subjective Opioid Withdrawal Scale (SOWS) | Baseline to day 7
  Change in pre- and post- intervention changes using SOWS
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely).
Positive and Negative Affect Scales (PANAS) | Baseline to day 7
  Change in severity of negative affect scores from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Opioid Craving Scale (OCS) | Baseline to day 14
  Change in pre- and post- intervention changes using OCS
  The Opioid Craving Scale is used to measure opioid craving. The scale consists of three items rated on a visual analogue scale from 0-10: (1) How much do you currently crave opiates? (rated from not at all to extremely), (2) In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates (rated from no desire to extremely strong), and (3) Please imagine yourself in the environment in which you previously used opiates. If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today? (rated from not at all to I'm sure I would use opiates).
Cocaine Craving Questionnaire-Brief (CCQ-Brief) | Baseline to day 14
  Change in pre- and post- intervention changes using CCQ-Brief
  The Cocaine Craving Questionnaire-Brief (CCQ-Brief) consists of 10 statements about the respondent's feelings and thoughts about using cocaine as her or she is completing the questionnaire (i.e., right now). This instrument allows investigators to obtain a reflection of the respondent's general cocaine craving.
Self-report instruments for Alcohol Craving | Baseline to day 14
  Change in pre- and post- intervention changes using self-report instruments for alcohol craving
  Administration of a single-item instrument on which the participant reports his or her level of subjective craving. These instruments include questions such as "How strong is your craving for alcohol?" or "How strong is your urge to drink?"
Subjective Opioid Withdrawal Scale (SOWS) | Baseline to day 14
  Change in pre- and post- intervention changes using SOWS
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely).
Positive and Negative Affect Scales (PANAS) | Baseline to day 14
  Change in severity of negative affect scores from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Opioid Craving Scale (OCS) | Baseline to Day 28
  Change in pre- and post- intervention changes using OCS
  The Opioid Craving Scale is used to measure opioid craving. The scale consists of three items rated on a visual analogue scale from 0-10: (1) How much do you currently crave opiates? (rated from not at all to extremely), (2) In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates (rated from no desire to extremely strong), and (3) Please imagine yourself in the environment in which you previously used opiates. If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today? (rated from not at all to I'm sure I would use opiates).
Cocaine Craving Questionnaire-Brief (CCQ-Brief) | Baseline to day 28
  Change in pre- and post- intervention changes using CCQ-Brief
  The Cocaine Craving Questionnaire-Brief (CCQ-Brief) consists of 10 statements about the respondent's feelings and thoughts about using cocaine as her or she is completing the questionnaire (i.e., right now). This instrument allows investigators to obtain a reflection of the respondent's general cocaine craving.
Self-report instruments for Alcohol Craving | Baseline to day 28
  Change in pre- and post- intervention changes using self-report instruments for alcohol craving
  Administration of a single-item instrument on which the participant reports his or her level of subjective craving. These instruments include questions such as "How strong is your craving for alcohol?" or "How strong is your urge to drink?"
Subjective Opioid Withdrawal Scale (SOWS) | Baseline to day 28
  Change in pre- and post- intervention changes using SOWS
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely).
Positive and Negative Affect Scales (PANAS) | Baseline to day 28
  Change in severity of negative affect scores from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Addiction Severity Index (ASI) | Baseline to day 28
  Monthly severity of opioid, stimulants and alcohol use using the ASI-modified
  The ASI is an assessment tool used to gauge the severity of a person's substance abuse and provides a comprehensive overview of a person's addiction-related issues. It addresses seven (7) main aspects of a person's behavior and environment. The areas assessed include medical status, employment and support, drug use, alcohol use, legal status, family/social status, and psychiatric status.
  The ASI substance abuse assessment uses the composite score to assign a severity rating. The ratings are based on a scale of 0 to 9 as follows:
  0-1: No imminent problem, treatment not indicated. 2-3: Slight problem; treatment may not be necessary. 4-5: Moderate problem, a treatment plan should be considered. 6-7: Considerable difficulty, begin a treatment plan. 8-9: Extreme problem, treatment is vital.
Opioid Craving Scale (OCS) | Baseline to 8 weeks
  Change in pre- and post- intervention changes using OCS
  The Opioid Craving Scale is used to measure opioid craving. The scale consists of three items rated on a visual analogue scale from 0-10: (1) How much do you currently crave opiates? (rated from not at all to extremely), (2) In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates (rated from no desire to extremely strong), and (3) Please imagine yourself in the environment in which you previously used opiates. If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today? (rated from not at all to I'm sure I would use opiates).
Cocaine Craving Questionnaire-Brief (CCQ-Brief) | Baseline to 8 weeks
  Change in pre- and post- intervention changes using CCQ-Brief
  The Cocaine Craving Questionnaire-Brief (CCQ-Brief) consists of 10 statements about the respondent's feelings and thoughts about using cocaine as her or she is completing the questionnaire (i.e., right now). This instrument allows investigators to obtain a reflection of the respondent's general cocaine craving.
Self-report instruments for Alcohol Craving | Baseline to 8 weeks
  Change in pre- and post- intervention changes using self-report instruments for alcohol craving
  Administration of a single-item instrument on which the participant reports his or her level of subjective craving. These instruments include questions such as "How strong is your craving for alcohol?" or "How strong is your urge to drink?"
Subjective Opioid Withdrawal Scale (SOWS) | Baseline to 8 weeks
  Change in pre- and post- intervention changes using SOWS
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely).
Positive and Negative Affect Scales (PANAS) | Baseline to 8 weeks
  Change in severity of negative affect scores from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Addiction Severity Index (ASI) | Baseline to 8 weeks
  Monthly severity of opioid, stimulants and alcohol use using the ASI-modified
  The ASI is an assessment tool used to gauge the severity of a person's substance abuse and provides a comprehensive overview of a person's addiction-related issues. It addresses seven (7) main aspects of a person's behavior and environment. The areas assessed include medical status, employment and support, drug use, alcohol use, legal status, family/social status, and psychiatric status.
  The ASI substance abuse assessment uses the composite score to assign a severity rating. The ratings are based on a scale of 0 to 9 as follows:
  0-1: No imminent problem, treatment not indicated. 2-3: Slight problem; treatment may not be necessary. 4-5: Moderate problem, a treatment plan should be considered. 6-7: Considerable difficulty, begin a treatment plan. 8-9: Extreme problem, treatment is vital.
Opioid Craving Scale (OCS) | Baseline to three months
  Change in pre- and post- intervention changes using OCS
  The Opioid Craving Scale is used to measure opioid craving. The scale consists of three items rated on a visual analogue scale from 0-10: (1) How much do you currently crave opiates? (rated from not at all to extremely), (2) In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates (rated from no desire to extremely strong), and (3) Please imagine yourself in the environment in which you previously used opiates. If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today? (rated from not at all to I'm sure I would use opiates).
Cocaine Craving Questionnaire-Brief (CCQ-Brief) | Baseline to three months
  Change in pre- and post- intervention changes using CCQ-Brief
  The Cocaine Craving Questionnaire-Brief (CCQ-Brief) consists of 10 statements about the respondent's feelings and thoughts about using cocaine as her or she is completing the questionnaire (i.e., right now). This instrument allows investigators to obtain a reflection of the respondent's general cocaine craving.
Self-report instruments for Alcohol Craving | Baseline to three months
  Change in pre- and post- intervention changes using self-report instruments for alcohol craving
  Administration of a single-item instrument on which the participant reports his or her level of subjective craving. These instruments include questions such as "How strong is your craving for alcohol?" or "How strong is your urge to drink?"
Subjective Opioid Withdrawal Scale (SOWS) | Baseline to three months
  Change in pre- and post- intervention changes using SOWS
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely).
Positive and Negative Affect Scales (PANAS) | Baseline to three months
  Change in severity of negative affect scores from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Addiction Severity Index (ASI) | Baseline to three months
  Monthly severity of opioid, stimulants and alcohol use using the ASI-modified
  The ASI is an assessment tool used to gauge the severity of a person's substance abuse and provides a comprehensive overview of a person's addiction-related issues. It addresses seven (7) main aspects of a person's behavior and environment. The areas assessed include medical status, employment and support, drug use, alcohol use, legal status, family/social status, and psychiatric status.
  The ASI substance abuse assessment uses the composite score to assign a severity rating. The ratings are based on a scale of 0 to 9 as follows:
  0-1: No imminent problem, treatment not indicated. 2-3: Slight problem; treatment may not be necessary. 4-5: Moderate problem, a treatment plan should be considered. 6-7: Considerable difficulty, begin a treatment plan. 8-9: Extreme problem, treatment is vital.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nwaokobia, Principal Investigator — Evon Medics LLC; Evaristus Nwulia, MD, Principal Investigator — Evon Medics LLC; Tanya Alim, MD, Principal Investigator — Howard University; Edwin Chapman, MD, Principal Investigator — Clinics of Dr. Edwin Chapman at MHDG; Marc Fishman, MD, Principal Investigator — Maryland Treatment Center
Locations (3):
- United States (3):
  - Clinics of Dr. Edwin Chapman @ MHDG, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Maryland Treatment Center, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No